CLINICAL TRIAL: NCT06845891
Title: Estudio clínico: Analisis de Control Glucemico y Satisfaccion Con un Cap Conectado en Pacientes Con dm Tipo 1
Brief Title: Clinical Study: Analysis of Glycemic Control and Satisfaction With a Connected Smart Cap in Patients With Type 1 Diabetes Mellitus
Acronym: CAPSDM1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fernando Sebastián Valles (Other)
Responsible Party: Sponsor-Investigator, Fernando Sebastián Valles, Medical doctor, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5350; 5350 (Registry Identifier: Estudio clínico: analisis de control glucemico y satisfaccion con un cap conectado en pacientes con DM tipo 1)
Record Dates: First submitted 2025-02-17; First posted 2025-02-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus; Type 1 Diabetes Mellitus (T1DM); Diabetes Management
Keywords: diabetes tecnhology; Type 1 diabetes; Smart cap; Time above range
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The healthcare provider will introduce the study to each individual with type 1 diabetes who meets the inclusion and exclusion criteria during routine medical visits. Subsequently, the research team will contact each participant and randomly assign the device. Given that the total study duration for each patient is two months, the study will conclude for each individual at their follow-up visit with the healthcare provider.
  Blinding will not be feasible for either participants or investigators, as the control group will not have access to the real-time data provided by the cap, which is linked to the digital application of the glucose monitoring sensor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Connected smart cap (Experimental): This arm will have access to the cap, which is connected to the digital application that records the timing of insulin injections and provides reminders in case of missed doses.
  Interventions: Device: CONNECTED SMART CAP
- cap disconnected (Active Comparator): This treatment arm will receive the cap without connectivity, thereby lacking access to the information provided by the digital application, including the timing of insulin injections, injection events, and reminder notifications.
  Interventions: Device: CONNECTED SMART CAP

INTERVENTIONS:
Device: CONNECTED SMART CAP — The intervention in this study consists of attaching a smart cap to the insulin pen of individuals with type 1 diabetes who use flash glucose monitoring and experience a time above range (TAR >180 mg/dL) for more than 25% of the time. This metric has been associated with diabetes-related complications, and the objective of this study is to determine whether this simple device could help reduce this underexplored parameter.

SUMMARY:
This clinical study evaluates the impact of the Cap INSULCLOCK device on glycemic control, treatment adherence, and patient satisfaction in adults with type 1 diabetes mellitus (T1DM). Despite advances in pharmacology and technology, a significant proportion of individuals with T1DM fail to achieve recommended glycemic targets, partly due to the complexity of insulin therapy and suboptimal adherence. Cap INSULCLOCK is a device that attaches to insulin pens, automatically recording injections and integrating data on glucose levels, insulin administration, food intake, and physical activity, with real-time Bluetooth transmission. Its use may enhance adherence and optimize metabolic control.

This study is a randomized, low-intervention clinical trial conducted at a single center, enrolling 42 patients, who will be randomized into two groups: one using the activated device and a control group using the device in a blinded mode. The primary objective is to assess differences in time above range (TAR >180 mg/dL) over the last 14 days of continuous glucose monitoring (CGM). Secondary objectives include evaluating HbA1c levels, time in range (TIR), frequency of hypoglycemic episodes, and patient satisfaction. Data will be analyzed using advanced statistical methods, and the intervention is expected to improve adherence, reduce glycemic variability, and enhance quality of life in individuals with T1DM

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older.
* Diagnosis of type 1 diabetes mellitus (T1DM).
* Users of flash continuous glucose monitoring (FGM) sensors with >70% of recorded data, including intake and insulin dose logs.
* Adequate therapeutic adherence, with no missed appointments in the past year.
* Time above range (TAR >180 mg/dL) >25%.
* Ability to provide informed consent to participate in the study.
* Access to technology for follow-up, including a smartphone with internet connectivity and compatibility with the Insulcloud app.

Exclusion Criteria:

* Current pregnancy.
* Severe acute illness.
* Exclusion criteria for the use of real-time continuous glucose monitoring (RT-CGM) systems as per the Framework Agreement of the Community of Madrid for RT-CGM use (SERMAS).
* Inability to provide informed consent or to meet the study requirements for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Time Above Range >180 mg/dL | 14 days
  Time Above Range (TAR) refers to the percentage of time that an individual's glucose levels exceed 180 mg/dL during a given period, in this case, the last 14 days as recorded by a continuous or flash glucose monitoring system. This metric reflects hyperglycemic burden and has been associated with an increased risk of diabetes-related complications. Clinical guidelines generally recommend keeping TAR below 25% to optimize glycemic control and reduce long-term adverse outcomes.

SECONDARY OUTCOMES:
Time in range (70 - 180 mg/dL), | 14 days
  Time in Range (TIR) refers to the percentage of time an individual's glucose levels remain within the target range of 70-180 mg/dL over the last 14 days, as recorded by a continuous or flash glucose monitoring system. TIR is a key glycemic metric reflecting overall glucose control, with higher percentages being associated with a lower risk of diabetes-related complications. Clinical guidelines recommend maintaining TIR above 70% as a primary therapeutic goal for individuals with diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to ethical and regulatory considerations regarding patient confidentiality

REFERENCES:
- [Derived] Sebastian-Valles F, Sager-La Ganga C, Justel Enriquez A, Jimenez Blanco S, Navas-Moreno V, Arranz Martin JA, Marazuela M. Analysis of glycaemic control and treatment satisfaction with a connected smart pen cap in adults with type 1 diabetes: a randomised, open-label, parallel-group trial. Diabetologia. 2026 Feb 3. doi: 10.1007/s00125-026-06674-w. Online ahead of print. PMID 41634174